CLINICAL TRIAL: NCT04716686
Title: Niraparib Monotherapy as Maintain and Recurrent Treatment of Endometrial Serous Carcinoma: A Multi-center, Open-label, Prospective Clinical Study
Brief Title: Niraparib Monotherapy as Maintain and Recurrent Treatment of Endometrial Serous Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Sun Yat-sen University (Other); Tongji Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Beihua Kong, professor, Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2306-914
Record Dates: First submitted 2020-12-09; First posted 2021-01-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Endometrial Carcinoma; Serous Carcinoma
Keywords: Endometrial Serous carcinoma; maintenance therapy; recurrent therapy; PARP inhibitor
MeSH Terms: conditions — Endometrial Neoplasms; Cystadenocarcinoma, Serous | interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niraparib as maintenance therapy for Endometrial Serous Carcinoma (Experimental): For patients with baseline weight ≥ 77 kg and baseline platelets ≥ 150000/uL, a starting dose of 300 mg QD will be given; other patients will be given a starting dose of 200 mg QD. One treatment cycle is 28 days; follow-up and evaluation will be conducted every 2 cycles until the disease progression or patients cannot tolerate.
  Interventions: Drug: Niraparib
- Niraparib as recurrent therapy for Endometrial Carcinoma (Experimental): For patients with baseline weight ≥ 77 kg and baseline platelets ≥ 150000/uL, a starting dose of 300 mg QD will be given; other patients will be given a starting dose of 200 mg QD. One treatment cycle is 28 days; follow-up and evaluation will be conducted every 2 cycles until the disease progression or patients cannot tolerate.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Patients received oral niraparib 200/300 mg QD and every cycle (28 days) thereafter until disease progression.

SUMMARY:
Endometrial Serous carcinoma (ESC) has similar molecular characteristics to high-grade serous ovarian carcinoma (HGSOC) and basal cell-like breast cancer, such as similar Chromosomal instability, somatic copy number variation profiles and somatic mutations. The clinical treatment of ESC also refers to the treatment model of HGSOC. The PARP inhibitor niraparib used in this study, which was approved by FDA for the maintenance treatment of adult patients with recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in complete or partial response to platinum-based chemotherapy on March 27, 2017.

The homologous recombination related gene mutations in total endometrial cancer accounted for 22%. Homologous Recombination Repair Defect (HRD) +ARID1A accounted for 48%, and 53% of endometrial cancer cell lines were sensitive to PARP inhibitors. The incidence of HRD in endometrial cancer with high copy number (the pathological type is mainly ESC) is 50%, suggesting potential clinical applications of PARP inhibitors for the treatment of ESC.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or above
* Histological confirmation of serous endometrial cancer or other types of endometrial cancer
* FIGO stage III-IV
* ESC Patients have received at least 6 cycles of first-line platinum containing chemotherapy after surgery and achieved CR, PR or SD; ESC patients have received platinum containing chemotherapy after the first relapse and achieved CR, PR or SD; these two types of patients are enrolled in cohort 1 and receive niraparib alone as maintenance therapy within 12 weeks after the last chemotherapy treatment.
* ESC Patients have received >2 lines of platinum containing chemotherapy and relapsed; patients with other types of endometrial cancer have received >2 lines of platinum containing chemotherapy and have BRCA mutation or be defined as HRD positive; these 2 types of patients are enrolled in cohort 2 and receive niraparib monotherapy.
* Radiotherapy or endocrine therapy history is allowed
* Cohort 1 life expectancy> 6 months; Cohort 2 life expectancy> 4 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Patients agreed to provide blood samples for testing BRCA status and HRR mutations.
* Patients agreed to provide formalin-fixed and paraffin-embedded tumor tissue samples for the detection of homologous recombination repair related genes (optional)
* Laboratory criteria are as follows:
* Neutrophil count ≥1500/µL;Platelets ≥100,000/µL;Hemoglobin ≥10g/dL;Serum creatinine ≤1.5 times of the upper limit, or creatinine clearance ≥60mL/min;Total bilirubin ≤1.5 times of the upper limit or direct bilirubin ≤1.0 times of the upper limit;AST and ALT ≤2.5 times of the upper limit, and must be ≤5 times of the upper limit of when liver metastasis exists.
* Patients of reproductive potential must have a negative urinary or serum pregnancy test when done and promise to take effective contraceptive measuresduring the period of the study; Or without potential fertility, defined as:
* Women who have undergone contraceptive operation(hysterectomy, bilateral oophorectomy or bilateral salpingectomy), or
* over 60 years old, or≥40 and <60 years of age, menopause for more than 12 months, and follicle-stimulating hormone test results are within the reference range of research institutions after menopause
* Willingness to sign a written informed consent document and follow the plan
* Any previous toxic and side effects of chemotherapy have recovered to ≤ CTCAE level 1 or baseline level, except for sensory neuropathy or hair loss with stable symptoms ≤ CTCAE level 2

Exclusion Criteria:

* Allergic to active or inactive ingredients of ZL-2306 (nirapali) or drugs with similar chemical structure to ZL-2306 (nirapali)
* Stage Ia(on invasion to myometrium)
* Symptomatic, uncontrollable brain metastases or pial metastases(No imaging scan is required); patients with spinal cord compression can still be considered for enrollment if they have received targeted therapy and have evidence of clinically SD for at least 28 days (patients with controlled central nervous system metastasis must have received radiotherapy or chemotherapy at least 1 month before and with no new symptoms related to central nervous system lesions or symptoms suggesting disease progression)
* Received surgery within 3 weeks before the start of the study, or any surgical effects that have not recovered.
* Received palliative radiotherapy with >20% bone marrow 1 week before enrollment
* Suffered from other aggressive cancers (except for fully treated basal or squamous cell skin cancer) within 2 years before enrollment
* Previously or currently diagnosed as myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Suffer from serious or uncontrollable diseases, including but not limited to:
* Uncontrollable nausea and vomiting, inability to swallow drugs, any gastrointestinal diseases that may interfere with drug absorption and metabolism
* Active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.
* Uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental disorders
* Immune deficiency (except for splenectomy)
* Any past or current disease, treatment or laboratory abnormality that may interfere with the results of the study, or be defined as not suitable for this study
* Receive platelet or red blood cell transfusion within 4 weeks before the start of the study.
* Pregnant or breastfeeding, or expect to become pregnant during the study.
* Have received any PARP inhibitor treatment previously.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS%（1 year） | assessed up to 12 months
  for maintenance therapy arm
Objective Response Rate (ORR) | assessed up to 30months]
  for maintenance therapy arm

SECONDARY OUTCOMES:
PFS%（2 year） | assessed up to 24 months
  for maintenance therapy am
Overall Survival (OS) | assessed up to 30 months
  for maintenance therapy am
Median PFS | assessed up to 30 months
  for recurrent therapy am
TEAEs | assessed up to 30 months
  for maintain and recurrent therapy arms

OTHER OUTCOMES:
PFS/ORR of Participants with BRCA+ or HRD+ | assessed up to 30 months
  for maintain / recurrent therapy arms

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Yoon JH, Yoo SC, Kim WY, Chang SJ, Chang KH, Ryu HS. Para-aortic lymphadenectomy in the management of preoperative grade 1 endometrial cancer confined to the uterine corpus. Ann Surg Oncol. 2010 Dec;17(12):3234-40. doi: 10.1245/s10434-010-1199-5. Epub 2010 Jun 29. PMID 20585865
- [Background] Kaelin WG Jr. The concept of synthetic lethality in the context of anticancer therapy. Nat Rev Cancer. 2005 Sep;5(9):689-98. doi: 10.1038/nrc1691. PMID 16110319
- [Background] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott CL, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Dougherty B, Orr M, Hodgson D, Barrett JC, Matulonis U. Olaparib maintenance therapy in patients with platinum-sensitive relapsed serous ovarian cancer: a preplanned retrospective analysis of outcomes by BRCA status in a randomised phase 2 trial. Lancet Oncol. 2014 Jul;15(8):852-61. doi: 10.1016/S1470-2045(14)70228-1. Epub 2014 May 31. PMID 24882434
- [Background] Kaufman B, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmana J, Mitchell G, Fried G, Stemmer SM, Hubert A, Rosengarten O, Steiner M, Loman N, Bowen K, Fielding A, Domchek SM. Olaparib monotherapy in patients with advanced cancer and a germline BRCA1/2 mutation. J Clin Oncol. 2015 Jan 20;33(3):244-50. doi: 10.1200/JCO.2014.56.2728. Epub 2014 Nov 3. PMID 25366685
- [Background] Watkins JA, Irshad S, Grigoriadis A, Tutt AN. Genomic scars as biomarkers of homologous recombination deficiency and drug response in breast and ovarian cancers. Breast Cancer Res. 2014 Jun 3;16(3):211. doi: 10.1186/bcr3670. PMID 25093514
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- See also: NCCN guidelines for ovarian cancer version 1 2019 — https://www.nccn.org/store/login/login.aspx?ReturnURL=https://www.nccn.org/professionals/physician_gls/pdf/ovarian.pdf